CLINICAL TRIAL: NCT05107167
Title: Electromagnetic Stimulation of the Phrenic Nerve to Generate Contraction of the Diaphragm in Anesthetized and Intubated Patients With Obesity - a Proof-of-concept Study
Brief Title: Electromagnetic Stimulation of the Phrenic Nerve of Intubated Patients With Obesity
Acronym: STIMIT-IA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Stimit AG (Industry)
Responsible Party: Principal Investigator, Stefan J Schaller, Deputy Clinical Director, Charite University, Berlin, Germany
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STIMIT-IA
Record Dates: First submitted 2021-10-26; First posted 2021-11-04 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-02

CONDITIONS: General Anaesthesia; Muscle Weakness
Keywords: VIDD; ICUAW; muscle weakness
MeSH Terms: conditions — Muscle Weakness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Electromagnetic stimulation (Experimental): Electromagnetic stimulation of the phrenic nerve.
  Interventions: Device: Electromagnetic stimulation

INTERVENTIONS:
Device: Electromagnetic stimulation — Electromagnetic stimulation of the phrenic nerve

SUMMARY:
Ventilator-induced diaphragmatic dysfunction is a common issue in critically ill patients. Muscle stimulation has shown to have beneficial effects in muscle groups on the extremities. A non-invasive way to stimulate the diaphragm would be the electromagnetic stimulation but it is currently unclear if that is feasible.

In this proof-of-concept trial the primary aim is to show that it is possible to induce a diaphragmatic contraction leading to an inspiration with a sufficient tidal volume via an external electromagnetic stimulation of the phrenic nerve in obese patients.

DETAILED DESCRIPTION:
During the time of first spontaneous breathing trial 60% of mechanically ventilated patients present with diaphragmatic weakness or also know as ventilator-induced diaphragmatic dysfunction (VIDD). The damage to the diaphragm in terms of muscle atrophy has been shown as early as 12 hours after initiation of mechanical ventilation. Recently, a correlation between diaphragmatic atrophy and mortality could be established.

Induction of diaphragmatic contractions via stimulation of the phrenic nerve would be a possible method to prevent or treat VIDD. A possible modality would be the non-invasive electromagnetic stimulation but feasibility has not been established.

In this proof-of-concept trial the primary aim is to show that it is possible to induce a diaphragmatic contraction leading to an inspiration with a sufficient tidal volume via an external electromagnetic stimulation of the phrenic nerve in obese patients

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* American Society of Anaesthesiologists Classification I or II
* Planned anesthesia with intubation
* Adipositas Grade II-III

Exclusion Criteria:

* Chronic lung disease
* Preexisting diaphragmatic weakness
* Neurologic disease with known motor weakness
* Paralysis of the phrenic nerve
* Contraindication for any movement in the cervical vertebrae
* Conditions that limit the movement of the diaphragm e.g. ascites, increased intraabdominal pressure.
* Inability to communicate in the official language
* Infections, lesions or stricture in the neck area
* Implanted cardiac devices e.g. pace maker, defibrillator, event recorder
* Implanted medical pumps e.g. left ventricular assist device
* Metal implants in the upper body
* Preganancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2021-12-14 (Actual); Primary Completion 2022-04-25 (Actual); Study Completion 2022-04-25 (Actual)

PRIMARY OUTCOMES:
1.Tidal volume generated by electromagentical stimulation of the phrenic nerve (ml) | approximately 15 minutes
  Mean tidal volume of 10 consecutively stimulations of the phrenic nerve

SECONDARY OUTCOMES:
Max inspiratory flow after stimulation | approximately 15 minutes
  The maximal air flow created in the duct following stimulation of the N. phrenicus (meter / second)
Abdominal extension maximum | approximately 15 minutes
  Extension of the abdomen in centimeter measured via abdominal belt
Air pressure during each breath | approximately 15 minutes
  Change in pressure in the duct from expiration to inspiration (mbar)
Diaphragmatic thickening fraction | approximately 15 minutes
  Diaphragmatic contractility measured by ultrasound after N. phrenicus stimulation
Feedback/Stimulation locus relation | approximately 15 minutes
  When the stimulation locus is changed according to protocol the change of the triggered tidal volume is measured in % to the original location
Latency between stimulation and feedback | approximately 15 minutes
  Time between start and end of the stimulation in seconds
Intensity/Contractility relation | approximately 15 minutes
  Correlation between the simulation intensity and the diaphragmatic contractility
Time to find the optimal stimulation point of the N. phrenicus | approximately 15 minutes
  Time between first successful N. phrenicus stimulation and identification of the optimal stimulation locus in seconds
Distance between anatomical landmarks and optimal stimulation locus | approximately 15 minutes
  Distance between anatomical landmarks and optimal stimulation locus
Reproducibility of stimulation answer | approximately 15 minutes
  Variation of stimulated tidal volumes and diaphragm contraction using mean and standard deviation of each stimulation intensity
Incidence of Adverse Events during stimulation | approximately 15 minutes
  Adverse Events elicited by the electromagnetic stimulation

CONTACTS AND LOCATIONS:
Overall Officials: Stefan J Schaller, Prof. Dr., Principal Investigator — Charité - Universitätsmedizin Berlin, Berlin, Germany
Locations (1):
- Charité - Univiversitätsmedizin Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data can be requested on reasonable scientific request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After publication of scientific manuscript.
Access Criteria: Deidentified data can be requested on reasonable scientific request.